CLINICAL TRIAL: NCT02120313
Title: Inpatient Versus Outpatient Rehabilitation Following Total Knee Arthroplasty
Brief Title: Inpatient Versus Outpatient Rehabilitation After TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Anett Mau-Moeller, M.A., University of Rostock
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESAR
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Total Knee Arthroplasty
Keywords: rehabilitation; total knee arthroplasty

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- inpatient rehabilitation (Active Comparator): After discharge, patients participate in daily physical therapy for 3 weeks in a rehabilitation hospital.
  Interventions: Other: inpatient rehabilitation
- outpatient rehabilitation (Experimental): After discharge, patients participate in daily physical therapy for 3 weeks in an outpatient rehabilitation center.
  Interventions: Other: outpatient rehabilitation

INTERVENTIONS:
Other: inpatient rehabilitation
  Arms: inpatient rehabilitation
Other: outpatient rehabilitation
  Arms: outpatient rehabilitation

SUMMARY:
The purpose of this study is to compare the effectiveness of inpatient and outpatient rehabilitation following total knee arthroplasty. No studies exist that have evaluated these two rehabilitation programmes in a specific orthopaedic patient population with a focus on motor performance. We hypothesized that patients participating in outpatient care tend to be physically more active than patients in the rehabilitation clinic, leading to the assumption that outpatient rehabilitation has superior functional outcomes compared to the inpatient standard-of-care therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients with knee osteoarthritis and scheduled for primary TKA
* age: 50-80

Exclusion Criteria:

* BMI > 40
* musculoskeletal and neurological disorders that limit physical function
* any planned further joint surgery within 6 months
* substantial pain or functional limitation which make the patients unable to perform study procedures

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-04; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
physical activity (number of steps) | during the first seven days of rehabilitation and 3 months post surgery (posttest)
  over a period of 7 days using activPAL activity recording system

SECONDARY OUTCOMES:
gait performance | posttest (3 months after surgery)
  spatio-temporal and temprophasic gait parameters
maximal active and passive knee joint range of motion | change from baseline (9 days after surgery) to posttest (3 months after surgery)
  digital long-arm goniometer
stair climbing performance | change from baseline (9 days after surgery) to posttest (3 months after surgery)
  stair climbing test
timed up and go performance | change from baseline (9 days after surgery) to posttest (3 months after surgery)
  timed up and go test
joint position sense | change from baseline (9 days after surgery) to posttest (3 months after surgery)
  The subjects' ability to actively reproduce a previously presented knee flexion angle (30° and 50° of knee Flexion)
knee pain | change from baseline (9 days after surgery) to posttest (3 months after surgery)
  visual analogue scale
knee joint swelling | change from baseline (9 days after surgery) to posttest (3 months after surgery)
  measurement of circumference
long-term Memory representation of the gait | change from baseline (9 days after surgery) to posttest (3 months after surgery)
  structural dimensional analysis of mental representation (SDA-M)

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Bergschmidt, MD, Study Chair — Department of Orthopedics, University Medicine Rostock; Wolfram Mittelmeier, MD, Study Director — Department of Orthopedics, University Medicine Rostock; Anett Mau-Moeller, M.A., Principal Investigator — Department of Orthopedics, University Medicine Rostock; Stephan Tohtz, MD, Principal Investigator — Klinik für Orthopädie und Unfallchirurgie, HELIOS Klinikum Emil von Behring GmbH; Martin Behrens, Principal Investigator — Department of Kinesiology, University of Rostock; Tino Stöckel, PhD, Principal Investigator — Department of Kinesiology, University of Rostock
Locations (1):
- Department of Orthopedics, University Medicine Rostock, Rostock, Germany

REFERENCES:
- See also: Stiftung Oskar Helene Heim — http://www.stiftung-ohh.de/